CLINICAL TRIAL: NCT03401905
Title: Comparison and Effects of Low and High Frequency Percutaneous Electrical Nerve Stimulation on Myofascial Chronic Neck Pain Patients.
Brief Title: Effects of Low Versus High Frequency Percutaneous Electrical Nerve Stimulation on Chronic Neck Pain Patients.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centro Universitario La Salle (Other)
Responsible Party: Principal Investigator, Jose Vicente Leon Hernandez, Principal investigator., Centro Universitario La Salle
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CSEULS-PI-115/2016
Record Dates: First submitted 2017-12-21; First posted 2018-01-17 (Actual); Last update posted 2018-05-09 (Actual); Status verified 2018-05

CONDITIONS: Neck Pain; Chronic Pain; Myofascial Pain Syndrome
Keywords: Percutaneous electrical nerve stimulation; Myofascial trigger point
MeSH Terms: conditions — Neck Pain; Chronic Pain; Myofascial Pain Syndromes

STUDY DESIGN:
Intervention Model Description: Double blind randomized control trial.
Who Masked: Participant, Outcomes Assessor
Masking Description: Randomized list that was only known by the therapist. Subjects do not know about the treatment they were receiving.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Low frequency (Experimental): Percutaneous electrical nerve stimulation with frequency of 2 Hz and 120 microseconds of pulse width will be applied.
  Interventions: Procedure: Low frequency
- High frequency (Active Comparator): Percutaneous electrical nerve stimulation with frequency of 120 Hz and 200 microseconds of pulse width will be applied.
  Interventions: Procedure: High frequency

INTERVENTIONS:
Procedure: Low frequency — A dry needling on trapezius muscle is performed, until two local twitch responses are obtained. The needle is kept inside the trigger point, as it will be the negative electrode, and an adhesive electrode will be added as the positive one. After that, a low frequency TENS is applied, at 2 Hz frequency and 120 microseconds of pulse width.
  Other Names: Low frequency group
  Arms: Low frequency
Procedure: High frequency — A dry needling on trapezius muscle is performed, until two local twitch responses are obtained. The needle is kept inside the trigger point, as it will be the negative electrode, and an adhesive electrode will be added as the positive one. After that, a high frequency TENS is applied, at 12o Hz frequency and 200 microseconds of pulse width.
  Other Names: High frequency group
  Arms: High frequency

SUMMARY:
Comparison between high and low frequency percutaneous electrical nerve stimulation as treatment of myofascial chronic neck pain. The main hypothesis is that low frequency treatment will have more hypoalgesic effects than high frequency, and low frequency effects will last longer.

ELIGIBILITY:
Inclusion Criteria:

* Neck pain of more than 6 months of evolution.
* Pain level of more than 30 millimeter on the VAS scale.
* Active myofascial frigger points on upper trapezius muscle.

Exclusion Criteria:

* Upper limb radiculopathy.
* Recent whiplash.
* Cervicogenic dizziness.
* Migraine.
* Previous cervical surgery.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2018-02-09 (Actual); Primary Completion 2018-04-09 (Actual); Study Completion 2018-04-09 (Actual)

PRIMARY OUTCOMES:
Pain | Changes on pain will be assessed during one month follow up. Baseline will be measured on the first day and one month later pain score will be reassessed.
  Subjective feeling expressed by subjects in the area of discomfort. It will be measured by a Visual Analogue Scale, meaning a score of 0 points/centimiters "no pain" and a score of 10 points/centimiters "unbearable pain".

SECONDARY OUTCOMES:
Pressure pain threshold | Changes on pain will be assessed during one month follow up. Baseline will be measured on the first day and one month later pain score will be reassessed.
  Minimal amount of pressure that induces pain. An algometer will be used to measure pressure pain threshold. Units will be kilograms per square centimeter. The higher the score is, the less sensitive the area will be.
Neck disability index. | Pre treatment at the beginning of the study and one month later, on the last of the follow up period.
  Ten items questionnaire designed to asses the level of pain and self-assessment of cervical disability. The NDI (Spanish version) is composed of 10 questions related to daily functional activities. NDI presents an acceptable reliability with an intraclass correlation coeffcient (ICC) ranging from 0.50 to 0.98. It has been proposed that the clinically important difference required for NDI is seven points.
kinesiofobia | Pre treatment at the beginning of the study and one month later, on the last of the follow up period.
  Eleven items questionnaire designed to asses pain-related fear. TSK-11, Spanish version.

CONTACTS AND LOCATIONS:
Overall Officials: Jose V León Hernández, PhD, Principal Investigator — CSEU La Salle
Locations (1):
- CSEU La Salle, Madrid, Spain

IPD SHARING:
Plan to Share IPD: No
Data collected will be used only for research objective. Once the trial have finished, data will be destroyed.